CLINICAL TRIAL: NCT02589964
Title: Probiotics in the Reduction of Antibiotic Associated Diarrhea and Clostridium Difficile in Pneumonia Patients Within a Community Teaching Hospital
Brief Title: Probiotics in the Reduction of Antibiotic Associated Diarrhea
Acronym: Probiotics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Jenni Steinbrunner, Research Specialist, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13085
Record Dates: First submitted 2015-04-13; First posted 2015-10-28 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Clostridium Difficile
Keywords: probiotics; antibiotic associated diarrhea; clostridium difficile
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Treatment will be initiated within 48 hours of the first antibiotic and will be administered twice a day for 20 days. The treatment is Florajen-3. The ingredients in Florajen-3 are:
  Lactobacillus acidophilus-over 7.5 billion Bifidobacterium lactis-over 6.0 billion Bifidobacterium longum-over 1.5 billion
  Interventions: Dietary Supplement: Florajen-3
- Placebo (Placebo Comparator): Placebo will be initiated within 48 hours of the first antibiotic and will be administered twice a day for 20 days. The ingredients in the placebo are:
  Rice maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Florajen-3 — The probiotic treatment is the experimental aspect of the study. Treatment will be initiated within 48 hours of the first antibiotic and will be administered twice a day for 20 days.
  Other Names: probiotic
  Arms: Probiotic
Other: Placebo — The placebo treatment is the experimental aspect of the study. Treatment will be initiated within 48 hours of the first antibiotic and will be administered twice a day for 20 days.
  Arms: Placebo

SUMMARY:
The study will evaluate the effectiveness of probiotic therapy in reducing the incidence of antibiotic associated diarrhea (AAD) and Clostridium difficile associated diarrhea (CDAD) in pneumonia patients.

DETAILED DESCRIPTION:
The study will include patients admitted to Good Samariatan Hospital and placed on the pneumonia order set. After obtaining consent, subjects will be randomized to the proboiotic or placebo group. Subjects will be followed for 21 days after starting the study treatment to determine critical outcomes such as incidence of antibiotic-associated diarrhea and C-Diff. Other outcomes include length of stay, healthcare costs, and death.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Good Samaritan Hospital
* Placed on pneumonia order set
* Age 18+

Exclusion Criteria:

* Patient with inadequate coherency to understand consent
* Active Diarrhea at admission
* Non-controlled intestinal disease
* Documented positive C. difficile infection within the 3 months before enrollment
* Antibiotic use at hospital admission
* Immunosuppressive therapy
* Pregnancy
* Allergic to ingredients in Florajen-3
* Allergic to ingredients in placebo
* Immunocompromised state including:
* HIV with a low CD4 count
* Active malignancy receiving chemotherapy
* Medications including long-term steroids (>2 weeks), and disease modifying biologic agents
* Acquired immune deficiency
* Unable to take oral medication
* Less than 4 doses of probiotic or placebo
* Taking probiotic in the past 30 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Antibiotic Associated Diarrhea | 21 days after starting study treatment
  Subjects will be asked to keep a diary for 20 days after starting study treatment and will be contacted by a nurse approximately 21 days after starting study treatment

SECONDARY OUTCOMES:
Length of stay | during hospitalization up to 4 weeks
Mortality | During hospitalization up to 4 weeks
Healthcare costs | During hospitalization up to 4 weeks
  Healthcare costs include direct costs during hospital stay (room, meds, procedures). This is obtained through the TriHealth Decision Support department.
Clostridium difficile | 21 days after initiating study treatment
  Data is obtained though a follow-up call to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Amita Buddhdev, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The study was closed due to poor recruitment, so there is no data to share.